CLINICAL TRIAL: NCT06677164
Title: Gluteus Maximus Strengthening Exercises Augmented by High-Intensity Laser Therapy in Patients With Chronic Plantar Fasciopathy
Brief Title: Gluteus Maximus Strengthening Exercises Augmented by High-Intensity Laser Therapy in Patients With Plantar Fasciopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, associate professor, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: physiotherapy 3
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fascia
Keywords: Plantar heel pain; obese; laser therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: High intensity laser therapy combined with Gluteus Maximus strengthening exercise (Experimental): patients will receive High intensity laser therapy combined with Gluteus Maximus strengthening exercise
  Interventions: Procedure: Gluteus Maximus strengthening exercise; Device: high-intensity laser therapy
- Active Comparator: High intensity laser therapy (Active Comparator): patients will receive High intensity laser therapy.
  Interventions: Device: high-intensity laser therapy

INTERVENTIONS:
Procedure: Gluteus Maximus strengthening exercise — Maximus strengthening exercise for eight weeks using weight progression tools either elastic band or sand weight by assuming two modes of exercises (clamshell exercise, prone hip extension) with stretching exercise (hamstring, gastrocnemius, soleus, and plantar fascia) 2 sessions per week for 8 weeks
  Arms: Experimental: High intensity laser therapy combined with Gluteus Maximus strengthening exercise
Device: high-intensity laser therapy — A 3-phase treatment program will be performed in each session on the plantar fascia area. Treatment of trigger points in phase 1 and 2 by using power of 9 watts, E2C mode for 6 minute of 2 phases. The draining and vascularization-promoting application involve the whole foot sole, starting from the heel area in phase three by using power of 9 watts, CW mode with energy of 100J/cm2.

SUMMARY:
Plantar heel pain is one of the most commonly encountered problems of the feet in adults [1]. It accounts for nearly 11%-15% of all foot symptoms, The purpose of this study was to investigate the effectiveness of high intensity laser therapy combined with gluteus Maximus strengthening exercise on pain, thickness of plantar fascia, and function of the foot.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral plantar heel pain with or without calcaneal spur for more than 3 months.
* Tenderness at the insertion of the plantar fascia
* BMI index will be from 25 up to 30
* Patient will wear silicone insole .
* Diagnosis of PF based on orthopedic referral

Exclusion Criteria:

* Patients with presence of foot deformity,
* systemic inflammatory arthritis disease,
* foot surgery, or
* plantar heel pain due to trauma,
* wound, or infection in the foot,
* received oral corticosteroids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 3 months
  Pressure algometry (kg/cm2). Pressure algometry will be performed on both affected and healthy feet
Plantar fascia thickness | 3 months
  by using Ultrasonography, in a longitudinal view of the tendon in both affected and healthy feet (mm). the normal plantar fascia thickness is less than 4 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No